CLINICAL TRIAL: NCT05933044
Title: A Retrospective Observational, Multi-Centre, Cohort Study to Understand Real-World Treatment Patterns and Clinical Outcomes of Adult Patients With Locally Advanced, Unresectable Non-Small Cell Lung Cancer (Stage III) in Canada
Brief Title: RELEVANCE - RWE Study in Unresectable Non-Small Cell Lung Cancer (Stage III) in Canada
Acronym: RELEVANCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00028
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: real-world evidence, treatment patterns, clinical outcomes, durvalumab, chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Durvalumab cohort: All stage III non-small cell lung cancer (NSCLC) patients who received durvalumab
  Interventions: Drug: Durvalumab
- Non-durvalumab cohort: All stage III non-small cell lung cancer (NSCLC) patients who did not receive durvalumab

INTERVENTIONS:
Drug: Durvalumab — Chemoradiotherapy plus durvalumab
  Other Names: Imfinzi
  Groups: Durvalumab cohort

SUMMARY:
In the RELEVANCE study, we will develop a scalable electronic medical report data capture platform to collect and analyse real-world data in the stage III NSCLC population in Canada across several Canadian cancer centres. Subsequent analyses will examine treatment patterns and clinical outcomes, including overall survival, for these patients, stratified by durvalumab regimen or non-durvalumab regimen during the time of the PACIFIC Patient Support Program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Patients must have histologically or cytologically documented diagnosis of NSCLC with a locally advanced, or locally recurrent (stage III) disease between November 1, 2017 and December 31, 2019 at the centre (Note: durvalumab uptake rate requires a secondary index date, such as initiation of CRT before availability of durvalumab in May 2018)

Exclusion Criteria:

* Patients treated with durvalumab in clinical studies prior to the start date
* Clinical trial patients where treatments received are blinded in the patient medical records

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with stage III NSCLC who received treatment at one of the participating clinical centres across Canada from November 1, 2017 until December 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | November 1, 2017 to August 31, 2022

SECONDARY OUTCOMES:
Rate and type of resection | November 1, 2017 to August 31, 2022
Treatments received including rates of concurrent chemoradiotherapy (cCRT) and sequential chemoradiotherapy (sCRT) use in unresectable disease | November 1, 2017 to August 31, 2022
Proportion of PACIFIC regimen initiation and uptake in patients who received CRT | November 1, 2017 to August 31, 2022
  Uptake of durvaluamab in patients who received CRT
Reasons for treatment discontinuation | November 1, 2017 to August 31, 2022
Time-to-treatment discontinuation | November 1, 2017 to August 31, 2022
Time to durvalumab initiation following CRT | November 1, 2017 to August 31, 2022
Rate and type of adverse events of special interest in the durvalumab cohort | November 1, 2017 to August 31, 2022

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - BC Cancer, Vancouver, British Columbia
  - Queen Elizabeth (QE) II Health Sciences Centre, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4191R00028&attachmentIdentifier=2b0cda25-fc2f-4415-865a-61e4f46e3d4b&fileName=AstraZeneca_RELEVANCE_CSR_Synopsis_v1_August_30-2023.pdf&versionIdentifier=